CLINICAL TRIAL: NCT01543178
Title: A Study to Assess Repeat Treatment Efficacy and Safety of Rifaximin 550 mg TID in Subjects With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: Irritable Bowel Syndrome With Diarrhea (IBS-D) Rifaximin Re-Treatment Study
Acronym: TARGET3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RFIB3053
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: IBS; IBS-D; IBS with diarrhea; Diarrhea; Irritable bowel syndrome with diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rifaximin open-label (Experimental): Subjects will receive open-label rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up. Responders will continue into Maintenance Phase 1 (treatment free). Nonresponders will withdraw from the study.
  Subjects who meet criteria for recurrence in Maintenance Phase 1 enter the double-blind period and are randomized 1:1 to receive rifaximin 550 mg or placebo.
  Interventions: Drug: open-label rifaximin
- Double-blind rifaximin (retreatment) (Experimental): Subjects in this arm receive rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up (first retreatment) followed by Maintenance Phase 2 (6 weeks [treatment free]) followed by a second retreatment with rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up.
  Interventions: Drug: open-label rifaximin; Drug: double-blind rifaximin
- Double-blind placebo (retreatment) (Placebo Comparator): Subjects in this arm receive placebo TID for 2 weeks with a 4-week treatment-free follow-up (first retreatment) followed by Maintenance Phase 2 (6 weeks [treatment free]) followed by a second retreatment with placebo TID for 2 weeks with a 4-week treatment-free follow-up.
  Interventions: Drug: open-label rifaximin; Drug: double-blind placebo

INTERVENTIONS:
Drug: open-label rifaximin — 550 mg three times a day (open-label)
  Other Names: rifaximin
Drug: double-blind placebo — 3 times a day (double-blind)
  Other Names: Placebo
  Arms: Double-blind placebo (retreatment)
Drug: double-blind rifaximin — 550 mg three times a day (double-blind)
  Other Names: rifaximin
  Arms: Double-blind rifaximin (retreatment)

SUMMARY:
This study will evaluate the effectiveness and safety of repeat treatment with rifaximin 550 mg three times a day in patients with IBS with diarrhea who respond to initial treatment of rifaximin 550 mg three times a day.

DETAILED DESCRIPTION:
It is important in chronic conditions to have information about how a product that is intended for short course administration in order to confer prolonged benefit should be administered beyond the first cycle of use once symptoms reappear. This Phase 3 study will evaluate the efficacy and safety of repeat treatment with rifaximin 550 mg three times daily (TID) for 14 days in subjects with IBS-D who respond to an initial treatment course with rifaximin 550 mg TID for 14 days.

This study consists of several treatment phases outlined below:

Screening/Treatment 1 Phase. Subjects will receive single-blind placebo TID for 7-13 days and answer daily IBS symptom-related questions.

Treatment 2 Phase. Eligible subjects will receive open-label rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up. Responders will continue into Maintenance Phase 1. Nonresponders will withdraw from the study.

Maintenance Phase 1. Subjects will continue the treatment-free follow-up period for up to 18 weeks until either: 1) they experience recurrence or 2) enrollment is met in the Treatment 3 Phase (Double Blind Repeat Treatment Phase). Subjects who do not meet recurrence criteria by the end of the Maintenance Phase 1 will withdraw from the study.

Treatment 3 Phase/ Double Blind Repeat Treatment Phase. Subjects who meet criteria for recurrence will be randomized 1:1 to receive either rifaximin 550 mg TID or placebo TID for 2 weeks with a 4-week treatment-free follow-up.

Primary efficacy analysis will be performed at the end of the Treatment 3 Phase (at Week 6 of the double-blind period).

Maintenance Phase 2. All subjects continued into an additional treatment-free follow-up period of up to 6 weeks (Maintenance Phase 2).

Treatment 4 Phase/Second Repeat Treatment Phase. Subjects will receive the same double-blind treatment as previously assigned in the Treatment 3 Phase for 2 weeks with a 4-week treatment-free follow-up.

A lactulose breath test sub-study will be conducted at select sites.

ELIGIBILITY:
Inclusion Criteria:

* IBS confirmed by Rome III diagnostic criteria.
* At least 18 years of age.
* Colonoscopy within the past 10 years to rule out inflammatory bowel disease; or flexible sigmoidoscopy if < 50 years of age or previous colonoscopy > 10 years prior.
* Willing to maintain a stable diet. including vitamins, supplements, and nutraceuticals.

Exclusion Criteria:

* Diabetes (Type 1 or 2).
* Lactose intolerance and not controlled by a lactose-free diet.
* Pregnant or planning to become pregnant or is lactating.
* History of HIV or hepatitis B or C.
* Participation in investigational study within past 30 days.
* Taking rifaximin or any other antibiotic within past 60 days.
* Unstable cardiovascular or pulmonary disease, with change in treatment in last 30 days due to worsening disease condition.
* History of GI surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2583 (Actual)
Dates: Start 2012-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Bortey, PhD, Study Director — Bausch Health Americas, Inc.
Locations (232):
- United States (229):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Dothan, Alabama
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Selma, Alabama
  - Chandler, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - North Little Rock, Arkansas
  - Sherwood, Arkansas
  - Anaheim, California
  - Artesia, California
  - Carlsbad, California
  - Chula Vista, California
  - Concord, California
  - Encinitas, California
  - Encino, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Huntington Beach, California
  - La Mesa, California
  - La Mirada, California
  - Laguna Hills, California
  - Lakewood, California
  - Lincoln, California
  - Lomita, California
  - Long Beach, California
  - Los Angeles, California
  - Madera, California
  - Mill Valley, California
  - Montebello, California
  - North Hollywood, California
  - Orange, California
  - Redlands, California
  - Sacramento, California
  - San Carlos, California
  - San Diego, California
  - Vista, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Lone Tree, Colorado
  - Bridgeport, Connecticut
  - Bristol, Connecticut
  - Danbury, Connecticut
  - Torrington, Connecticut
  - Boca Raton, Florida
  - Boynton Beach, Florida
  - Brandon, Florida
  - Clearwater, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Hollywood, Florida
  - Jupiter, Florida
  - Kissimmee, Florida
  - Lake Worth, Florida
  - Largo, Florida
  - Lauderdale Lakes, Florida
  - Maitland, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - Naples, Florida
  - Orange Park, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Plant City, Florida
  - Pompano Beach, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - Seminole, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Wellington, Florida
  - West Palm Beach, Florida
  - Winter Haven, Florida
  - Winter Park, Florida
  - Zephyrhills, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Augusta, Georgia
  - Columbus, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Norcross, Georgia
  - Boise, Idaho
  - Hayden Lake, Idaho
  - Idaho Falls, Idaho
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Evanston, Illinois
  - Oak Lawn, Illinois
  - Elkhart, Indiana
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Mishawaka, Indiana
  - Clive, Iowa
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Bowling Green, Kentucky
  - Crestview Hills, Kentucky
  - Hebron, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Hollywood, Maryland
  - Boston, Massachusetts
  - Brockton, Massachusetts
  - Marlborough, Massachusetts
  - Watertown, Massachusetts
  - Ann Arbor, Michigan
  - Kalamazoo, Michigan
  - Saginaw, Michigan
  - Wyoming, Michigan
  - Jackson, Mississippi
  - Ocean Springs, Mississippi
  - Kansas City, Missouri
  - Lee's Summit, Missouri
  - Mexico, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Bellevue, Nebraska
  - Fremont, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Reno, Nevada
  - Lebanon, New Hampshire
  - Newington, New Hampshire
  - Haddon Heights, New Jersey
  - Marlton, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Great Neck, New York
  - Hollis, New York
  - Mineola, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Asheboro, North Carolina
  - Asheville, North Carolina
  - Boone, North Carolina
  - Cary, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - High Point, North Carolina
  - Kinston, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Groveport, Ohio
  - Kettering, Ohio
  - Mentor, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Downingtown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - Sayre, Pennsylvania
  - East Providence, Rhode Island
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Fort Mill, South Carolina
  - Gaffney, South Carolina
  - Greer, South Carolina
  - Brentwood, Tennessee
  - Bristol, Tennessee
  - Chattanooga, Tennessee
  - Franklin, Tennessee
  - Germantown, Tennessee
  - Hermitage, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - Odessa, Texas
  - Pasadena, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Sealy, Texas
  - Southlake, Texas
  - Tyler, Texas
  - Bountiful, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Danville, Virginia
  - Fairfax, Virginia
  - Richmond, Virginia
  - Suffolk, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Germany (2):
  - Berlin
  - Hamburg
- Manchester, United Kingdom

REFERENCES:
- [Derived] Lacy BE, Chang L, Rao SSC, Heimanson Z, Sayuk GS. Rifaximin Treatment for Individual and Multiple Symptoms of Irritable Bowel Syndrome With Diarrhea: An Analysis Using New End Points. Clin Ther. 2023 Mar;45(3):198-209. doi: 10.1016/j.clinthera.2023.01.010. Epub 2023 Mar 14. PMID 36922331
- [Derived] Fodor AA, Pimentel M, Chey WD, Lembo A, Golden PL, Israel RJ, Carroll IM. Rifaximin is associated with modest, transient decreases in multiple taxa in the gut microbiota of patients with diarrhoea-predominant irritable bowel syndrome. Gut Microbes. 2019;10(1):22-33. doi: 10.1080/19490976.2018.1460013. Epub 2018 Jul 18. PMID 29708822
- [Derived] Cash BD, Pimentel M, Rao SSC, Weinstock L, Chang L, Heimanson Z, Lembo A. Repeat treatment with rifaximin improves irritable bowel syndrome-related quality of life: a secondary analysis of a randomized, double-blind, placebo-controlled trial. Therap Adv Gastroenterol. 2017 Sep;10(9):689-699. doi: 10.1177/1756283X17726087. Epub 2017 Sep 11. PMID 28932270
- [Derived] Pimentel M, Cash BD, Lembo A, Wolf RA, Israel RJ, Schoenfeld P. Repeat Rifaximin for Irritable Bowel Syndrome: No Clinically Significant Changes in Stool Microbial Antibiotic Sensitivity. Dig Dis Sci. 2017 Sep;62(9):2455-2463. doi: 10.1007/s10620-017-4598-7. Epub 2017 Jun 6. PMID 28589238
- [Derived] DuPont HL, Wolf RA, Israel RJ, Pimentel M. Antimicrobial Susceptibility of Staphylococcus Isolates from the Skin of Patients with Diarrhea-Predominant Irritable Bowel Syndrome Treated with Repeat Courses of Rifaximin. Antimicrob Agents Chemother. 2016 Dec 27;61(1):e02165-16. doi: 10.1128/AAC.02165-16. Print 2017 Jan. No abstract available. PMID 27795384
- [Derived] Lembo A, Pimentel M, Rao SS, Schoenfeld P, Cash B, Weinstock LB, Paterson C, Bortey E, Forbes WP. Repeat Treatment With Rifaximin Is Safe and Effective in Patients With Diarrhea-Predominant Irritable Bowel Syndrome. Gastroenterology. 2016 Dec;151(6):1113-1121. doi: 10.1053/j.gastro.2016.08.003. Epub 2016 Aug 13. PMID 27528177

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The screening phase included a 10 (±3) day run-in treatment period, during which subjects received single-blind placebo and completed a daily IBS symptom diary. Subjects who had active symptoms of IBS with diarrhea, and satisfied other entry criteria, entered the open-label period of study.
Groups:
- Open-label Rifaximin: Subjects received open-label rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up. Responders continued into Maintenance Phase 1 (treatment free). Nonresponders withdrew from the study.
  Of the 2583 subjects in this group, 636 eventually met criteria for recurrence in Maintenance Phase 1, entered the double-blind period, and were randomized 1:1 to receive rifaximin 550 mg or placebo.
- Double-blind Rifaximin (Retreatment): The 328 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the rifaximin group for the double-blind retreatment period. For participant flow during the open-label period, these subjects are included in the 2583 subjects in the open-label rifaximin group.
- Double-blind Placebo (Retreatment): The 308 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the placebo group for the double-blind retreatment period. For participant flow during the open-label period, these subjects are included in the 2583 subjects in the open-label rifaximin group.
Period: Open-label Period
Arm/Group | Open-label Rifaximin | Double-blind Rifaximin (Retreatment) | Double-blind Placebo (Retreatment)
Started | 2583 (2583 subjects entered the open-label period, but 4 received no rifaximin; 2579 received rifaximin.) | 0 (The double-blind rifaximin arm/group is not applicable to the open-label period.) | 0 (The double-blind placebo arm/group is not applicable to the open-label period.)
Completed | 636 | 0 | 0
Not Completed | 1947 | 0 | 0
Period: Double-blind Period
Arm/Group | Open-label Rifaximin | Double-blind Rifaximin (Retreatment) | Double-blind Placebo (Retreatment)
Started | 0 (The open-label rifaximin arm/group is not applicable to the double-blind period.) | 328 (636 subjects had recurrence in open-label period; 328 randomized to rifaximin.) | 308 (636 subjects had recurrence in open-label period; 308 randomized to placebo.)
Completed | 0 | 284 (295 completed 1st double-blind retreatment and 284 completed 2nd double-blind retreatment.) | 271 (283 completed 1st double-blind retreatment and 271 completed 2nd double-blind retreatment.)
Not Completed | 0 | 44 | 37

BASELINE CHARACTERISTICS:
Population: Baseline results were summarized for the safety population, defined as patients who received at least 1 dose of study drug. Results are presented for patients in the open-label period only (1943) and for patients who eventually were randomized to rifaximin (329) or placebo (308) (ie, participated in both open-label and double-blind periods).
Groups:
- Open-label Rifaximin Only: The 1943 subjects in this group did not continue into the double-blind period of the study. Open-label treatment was rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up.
- Double-blind Rifaximin (Retreatment): The 328 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the rifaximin group for the double-blind retreatment period.
- Double-blind Placebo (Retreatment): The 308 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the placebo group for the double-blind retreatment period.
- Total: Total of all reporting groups
Arm/Group | Open-label Rifaximin Only | Double-blind Rifaximin (Retreatment) | Double-blind Placebo (Retreatment) | Total
Number analyzed (Participants) | 1943 | 328 | 308 | 2579
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 0 | 1 | 9
  Between 18 and 65 years | 1763 | 289 | 278 | 2330
  >=65 years | 172 | 39 | 29 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (13.5) | 47.9 (14.2) | 45.6 (13.8) | 46.4 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1319 | 222 | 219 | 1760
  Male | 624 | 106 | 89 | 819

OUTCOME MEASURES:

1. Primary Outcome: Repeat Treatment Responders
Description: Subjects who respond to repeat treatment in both IBS-related abdominal pain and stool consistency. The proportion of patients who responded to repeat treatment during the first double-blind repeat treatment phase is presented. Response is defined as improvement from baseline in abdominal pain AND reduction from baseline in diarrhea.
Time Frame: 4-week treatment-free follow-up in double-blind repeat treatment phase.
Population: Intent-to-treat population, defined as patients who received ≥ 1 dose of study drug in the double-blind period.
Measure: Number; unit: percentage of patients
Groups:
- Double-blind Rifaximin (Retreatment): The 328 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the rifaximin group for the double-blind retreatment period.
  During the double-blind period, subjects in this arm received rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up (first retreatment) followed by Maintenance Phase 2 (6 weeks [treatment free]) followed by a second retreatment with rifaximin.
- Double-blind Placebo (Retreatment): The 308 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the placebo group for the double-blind retreatment period.
  During the double-blind period, subjects in this arm received placebo TID for 2 weeks with a 4-week treatment-free follow-up (first retreatment) followed by Maintenance Phase 2 (6 weeks [treatment free]) followed by a second retreatment with placebo.
Arm/Group | Double-blind Rifaximin (Retreatment) | Double-blind Placebo (Retreatment)
Number analyzed (Participants) | 328 | 308
percentage of patients | 32.6 | 25.0
Statistical Analysis 1: Comparison: Double-blind Rifaximin (Retreatment) vs Double-blind Placebo (Retreatment); A worst case analysis was performed, in which patients with < 4 days of IBS symptom data in a given week were considered as non-responders for that week; Test type: Superiority or Other; p = 0.0232, Cochran-Mantel-Haenszel — The a priori threshold for statistical significance was p < 0.05; The Cochran-Mantel-Haenszel method was adjusted for analysis center and time to recurrence during Maintenance Phase 1

ADVERSE EVENTS:
Time Frame: Up to 24 weeks for the open-label period. Up to 18 weeks for the double-blind period.
Description: The tables below present serious adverse events and other adverse events that were reported during treatment with study drug and during off-treatment follow-up and maintenance phases. Non-systematic (patient reports) and systematic methods (investigator examinations and laboratory tests) were used to collect adverse events.
Groups:
- Total Open-label Experience: This group includes all 2579 subjects who received rifaximin the open-label period.
  Open-label experience is shown here.
- Double-blind Retreatment Experience - Rifaximin Group: The 328 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the rifaximin group for the double-blind retreatment period.
  During the double-blind period, subjects in this arm received rifaximin 550 mg TID for 2 weeks with a 4-week treatment-free follow-up (first retreatment) followed by Maintenance Phase 2 (6 weeks [treatment free]) followed by a second retreatment with rifaximin.
  Double-blind experience is shown here.
- Double-blind Retreatment Experience - Placebo Group: The 308 subjects in this group received rifaximin in the open-label period, eventually met criteria for recurrence and were randomized to the placebo group for the double-blind retreatment period.
  During the double-blind period, subjects in this arm received placebo TID for 2 weeks with a 4-week treatment-free follow-up (first retreatment) followed by Maintenance Phase 2 (6 weeks [treatment free]) followed by a second retreatment with placebo.
  Double-blind experience is shown here.
Arm/Group | Total Open-label Experience | Double-blind Retreatment Experience - Rifaximin Group | Double-blind Retreatment Experience - Placebo Group
Serious Adverse Events (participants affected / at risk) | 28/2579 | 4/328 | 4/308
Other Adverse Events (participants affected / at risk) | 198/2579 | 74/328 | 69/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Open-label Experience (N=2579) | Double-blind Retreatment Experience - Rifaximin Group (N=328) | Double-blind Retreatment Experience - Placebo Group (N=308)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 4 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Open-label Experience (N=2579) | Double-blind Retreatment Experience - Rifaximin Group (N=328) | Double-blind Retreatment Experience - Placebo Group (N=308)
Diarrhoea (Gastrointestinal disorders) | 20 | 7 | 3
Nausea (Gastrointestinal disorders) | 52 | 12 | 7
Vomiting (Gastrointestinal disorders) | 24 | 2 | 5
Bronchitis (Infections and infestations) | 15 | 9 | 5
Nasopharyngitis (Infections and infestations) | 36 | 10 | 9
Influenza (Infections and infestations) | 33 | 7 | 2
Sinusitis (Infections and infestations) | 34 | 7 | 7
Upper respiratory tract infection (Infections and infestations) | 41 | 12 | 8
Urinary tract infection (Infections and infestations) | 35 | 11 | 15
Alanine aminotransferase increased (Investigations) | 24 | 9 | 4
Aspartate aminotransferase increased (Investigations) | 24 | 7 | 4
Blood creatine phosphokinase increased (Investigations) | 31 | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 3 | 8
Headache (Nervous system disorders) | 42 | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days